CLINICAL TRIAL: NCT04987775
Title: Mechanisms of Oxidative Stress During N-Acetyl Cysteine (NAC) Supplementation in Veterans With Gulf War Illness (GWI)
Brief Title: GWICTIC: NAC Mechanistic Study in Gulf War Veterans
Acronym: NAC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: RTI International (Other); Boston University (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWICTIC-NAC
Record Dates: First submitted 2021-06-07; First posted 2021-08-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Gulf War Syndrome
Keywords: CNS Recovery; N-Acetyl Cysteine (NAC); Gulf War Illness; Placebo
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Participants enrolled will be randomized into one of two arms: NAC or Placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-Acetyl Cysteine (NAC) (Active Comparator): Participants who are randomized to the intervention arm will receive N-Acetyl-L-Cysteine (Free-Form/NAC) 900mg two times a day for 8 weeks after the initiation of the first dose of study drug.
  Interventions: Drug: N-Acetyl Cysteine
- Placebo (Placebo Comparator): Participants who are randomized to the placebo arm will take matching placebo two times a day for 8 weeks after the initiation of the first dose of study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetyl Cysteine — 900mg 2x daily
  Other Names: NAC
  Arms: N-Acetyl Cysteine (NAC)
Drug: Placebo — Matching placebo bid
  Other Names: NAC Placebo
  Arms: Placebo

SUMMARY:
This mechanistic study will test if NAC affects chronic oxidative stress and depletion of antioxidants in GWI participants. Blood specimen collection and neuroimaging will be used to determine whether NAC affects serum glutathione (GSH) concentration and oxidative stress in the CNS when compared to placebo.

DETAILED DESCRIPTION:
During the 1990-91 Gulf War (GW), military personnel were exposed to numerous chemical and environmental agents during deployment including spraying of pesticides, petroleum combustion products, and nerve gas. Exposure to these chemical and environmental agents can damage cell function and more specifically, mitochondrial function, which negatively affects energy production and can lead to oxidative stress and neuroinflammation. Animal models using similar exposures have documented this in the central nervous system (CNS) compartment. This disruption in mitochondrial function and energy production is likely tied to resulting symptoms of Gulf War Illness (GWI) including fatigue, headaches, joint and muscle pain, gastrointestinal and sleep disturbances, neurologic and neuropsychological symptoms, respiratory issues, and cardiovascular problems.

The Gulf War Illness Clinical Trials and Interventions Consortium (GWICTIC) plans to evaluate N-Acetyl Cysteine (NAC) as a promising approach to help the CNS recover from chronic oxidative stress and depletion of antioxidants. The Congressionally Directed Medical Research Program's (CDMRP's) two Gulf War Illness Consortiums (GWICs) and others have added to the growing evidence of the role of CNS oxidative stress and neuroinflammation in symptoms of GWI, yet there is little definitive work on the delivery of antioxidants to the CNS environment. In this mechanistic study, we aim to determine if NAC has the ability to target mitochondrial dysfunction and reverse oxidative stress in the CNS. Based on our early experiences with antioxidants in GWI and other complex disease states along with the proven record of NAC in reducing glutathione (GSH) deficits, it is possible that this antioxidant will help to restore mitochondrial function and provide a more targeted approach to improve outcomes in Veterans with GWI.

ELIGIBILITY:
Inclusion Criteria:

* 47 to 70 years
* Served in the Gulf War Theater for any period between August 1990 and July 1991.
* Meets modified Kansas case definition criteria for Gulf War Illness. The modified Kansas definition includes the following:

  1. Allowance of normal illness of aging, such as hypertension and diabetes, if the conditions are treated and are in demonstrable stable and normal ranges at the time of screening and assessment.
  2. Allowance of stable comorbid conditions such as Post Traumatic Stress Disorder (PTSD), Major Depressive Disorder (MDD), and mild Traumatic Brain Injury (mTBI) that have not required hospitalization in the 2 years prior to recruitment. Severe TBI is excluded.
* Able to provide written consent to the study
* Agrees to participate in follow-up visits.

Exclusion Criteria:

* Self-report of current treated or untreated major depression with psychotic or melancholic features (as determined by self-report and Hamilton Depression Inventory (Ham-D)), schizophrenia, bipolar disorder, delusional disorders, dementias of any type, or a history of central nervous system (CNS) disorders that may affect cognitive function (e.g., epilepsy, stroke, brain tumor, multiple sclerosis, Parkinson's Disease, Alzheimer's disease), or alcoholism or drug abuse
* Severe claustrophobia or serious difficulty being in an MRI scanner or other enclosed space (MRS substudy only)
* Presence of ferrous implanted medical devices or metal fragments or objects that are embedded under the skin (MRS substudy only)
* Current heavy alcohol or tobacco use (self-report). Alcohol consumption not to exceed approximately 15 drinks per week (with a drink defined as 12 oz beer, 5 oz wine, or 1.5 oz distilled spirits) and tobacco use not to exceed 20 cigarettes (or equivalent) per day.
* Chronic active infections such as HIV, Hepatitis B Virus (HBV), and Hepatitis C Virus (HCV) (self-report or antibody titer)
* Renal disease (self-report or laboratory results: renal insufficiency with serum creatinine > 2.0 mg/dL)
* Liver disease (self-report or laboratory results: hepatic insufficiency (bilirubin >2.5mg/dL or transaminases > 3 times the upper limits of normal)
* Uncontrolled diabetes (HgbA1c > 7.5) without adequate medical care. Individuals with HgbA1c > 7.5 will be reviewed and judged by the PI or delegate; if potential participant has adequate medical care to manage diabetes, enrollment is allowed; otherwise HgbA1c > 7.5 is exclusionary
* Diagnosed vascular disease (including congestive heart failure)
* Diagnosed bleeding disorders or use of blood-thinning medications
* Receipt of stavudine or didanosine for more than 7 days within 30 days prior to screening
* Currently have exclusionary diagnoses that could reasonably explain the symptoms of their fatiguing illness and their severity
* Are scheduled for a surgery during the period of study participation or had surgery within 6 weeks prior to screening
* Pregnant (women only)

Prohibited Concomitant or Prior Therapies

* Currently on dialysis
* Previous or current receipt of any antiviral medication, such as pegylated interferon, ribavirin, entecavir, tenofovir, or didanosine for more than 7 days within 30 days prior to screening
* Participating in another interventional (including social-behavioral therapy) clinical trial of an investigational therapy within 6 weeks prior to consent, or planning to participate in another interventional clinical trial of an investigational therapy during the course of this study
* Any herbal medicine within 30 days prior to consent and screening blood draw

Ages: 47 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assess glutathione levels | Baseline to 8 weeks
  Change in glutathione levels after NAC supplementation compared to placebo in participants with gulf war illness (GWI)

SECONDARY OUTCOMES:
Change in glutathione levels | Baseline to 8 Weeks
  Measure the change of brain glutathione levels with magnetic resonance spectroscopy (MRS) in a subset of both arms of study at baseline and 8 weeks.
Change in number of participants with treatment-related adverse events | Baseline to 16 Weeks
  Change in number of participants with treatment-related adverse events from baseline to 16 weeks during the intervention period as assessed by a safety questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Klimas, MD, Principal Investigator — Nova Southeastern Univeristy
Locations (7):
- United States (7):
  - VA Palo Alto Health Care System War Related Illness and Injury Study Center, Palo Alto, California
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Boston University Medical School, Boston, Massachusetts
  - VA New Jersey Health Care System War Related Illness and Injury Study Center, East Orange, New Jersey
  - Weill Cornell Medical College, New York, New York
  - RTI International, Durham, North Carolina
  - Michael E. DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
The plan is to release primary results from the study. Data are the property of Nova Southeastern University, but data and publication thereof will not be unduly withheld.